CLINICAL TRIAL: NCT03180580
Title: Feasibility and Acceptability of Implementing School Based "Healthy Eating and Active Living" Intervention to Control Overweight and Obesity Among Children in Urban Area in Bangladesh
Brief Title: School Based Childhood Obesity Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: The University of Queensland (Other); University of California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR-15057
Record Dates: First submitted 2016-09-08; First posted 2017-06-08 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2017-06

CONDITIONS: Overweight and Obesity
Keywords: Childhood, Overweight, Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HEAL guideline+ Healthy Tiffin box (Experimental): HEAL guideline+ Healthy Tiffin box intervention arm will receive a culturally appropriate healthy eating and active living messages including a specially designed healthy tiffin box to practice healthy eating. HEAL guideline+ Healthy Tiffin box is a combination of intervention to promote healthy eating and physical activity behavior as well as improve the practice.
  HEAL guideline-Healthy Eating and Active Living (HEAL) Guideline. A complete intervention guideline for promoting healthy dietary pattern and physical activity.
  Healthy Tiffin box- A five chamber snack box that will help to contain food stuffs from all 5 major food groups eg; grain, meat/fish foods, vegetables, fruits and milk or milk products. This box will help to practice healthy eating behaviors.
  Interventions: Behavioral: HEAL guideline and healthy tiffin box intervention

INTERVENTIONS:
Behavioral: HEAL guideline and healthy tiffin box intervention — Healthy Eating and Active Living (HEAL) guideline and healthy tiffin box intervention is a combination of intervention to promote healthy eating behavior and improve physical activity level of school going children. The guideline was developed to deliver healthy lifestyle message encouraging healthy dietary habit and physical activity pattern in order to control childhood overweight and obesity. Investigators was designed a "Healthy Tiffin Box" for children that contained five different compartments of various sizes for stuffing with five different food types in order to ensure healthy balanced diet including low carbohydrate, moderate protein, low fat and high vitamin. We also provided with a recommended physical activity list for children.

SUMMARY:
In Bangladesh, the prevalence of overweight and obesity among children varies from less than 1% to 17.9% based on different reference standard. In 2014 school based country wide study has been demonstrated that among children (6-15 years of age), 9.6% were overweight and 3.5% children were obese. Childhood obesity is getting increasing attention due to its association with adult obesity and increased risk of co morbidities in adulthood. Childhood obesity is known to be an independent risk factor for adult obesity and once a child is obese, it is difficult to reverse through interventions. This suggests an urgent need to address overweight and obesity levels in childhood. The increasing trend of childhood obesity suggests urgent solution of the problem. There is no evidence of intervention for childhood overweight and obesity exists in Bangladesh. This feasibility study will be able to generate evidence for overcoming this upcoming epidemic in resource poor setting. If the proposed study will be able to address its objective that will create a possibility for developing a large cluster randomized trial in low resource setting like Bangladesh. This study will also give opportunity to our policy makers for advocating to the government of Bangladesh for adopting an obesity control policy for children.

The aim of the study is to develop a school based healthy eating and active lifestyles module and assess feasibility and acceptability of the guideline in school setting.

Outcome measures/variables:

Healthy Eating and Active Living intervention material (Guideline, Tiffin box) Perception of children, parents and policy makers regarding obesogenic behavior Acceptance of children, parents and policy makers regarding planned intervention.

Facilitators and barriers of Healthy Eating and Active Living.

DETAILED DESCRIPTION:
Study Setting:

The investigators were purposively selected four wards with the highest prevalence of obesity out of 30 wards that were surveyed in the previous study (PR-13024) conducted by Centre for control of chronic diseases (CCCD), icddr,b. Investigators were obtained the list of schools from city corporation head office for the 4 selected wards. Investigators were randomly selected 2 English medium and 2 Bengali medium schools from the available list. Investigators were included only those schools who will give us a letter of supports for their voluntary participation in the research project. We were followed the available list of both Bengali and English medium schools collected from City Corporation. If any school disagrees to participate in the research, we were approached next available school in the list and selected following a letter of supports.

With supports of the school authority, investigators were assessed BMI of all children in Grade 3 (aged 7-8 years) up to Grade 9 (aged 13-14 years) in order to make a list of those children who will have a higher than normal BMI. Investigators were randomly selected 3 children from that list from each grade and obtain parental consent to recruit them. Investigators were additionally obtained assent for children 11-14 years of age. A written voluntary consent was provided to parents describing the study purpose, objectives and methodology prior to obtaining consent of the parents and get permission to recruit their child participate in the study. Thus investigators were recruited 27 children from one school and a total of 108 children were selected from 4 schools for inviting to participate in the intervention.

Study Design:

The study was adopted both of quantitative and qualitative designs. Investigators were conduct secondary analysis to achieve specific aim 1 using data on diet and physical activity pattern from previously conducted study by Centre for Control of Chronic Diseases (CCCD) in 2013 in 7 divisional cities in Bangladesh. For achieving aims 2, and 3 we were adopted qualitative methods.

To achieve specific aim 1, investigators were performed secondary data analysis to determine the usual dietary and physical activity pattern of the children. Investigators were analyzed data on childhood dietary pattern following food frequency questionnaire and food preference were also be calculated. There were 20 food groups for listing food preference that has been collected through 7 days recall method. These food groups were analyzed for children's food preference by rating 'preferred' and 'not preferred' as well as frequency of consumption within 24 hours and last 7 days. Thus we were determined the dietary patterns of children 5-18 years of age with normal BMI, high BMI and low-BMI which has already been defined in the study by following the International Obesity Task Force (IOTF) guideline. In order to develop healthy eating guideline, we were developed a dietary guideline that would be suitable for children with normal weight, and make adjustment in the dietary pattern for underweight and overweight children. We will determine appropriate portion size of carbohydrates, proteins, fats, vitamins and minerals required for a balanced nutritional supply for different ages. The total daily calorie intake should comprise of: Fat - 30-35%, Protein - 15% and Carbohydrates - 50-55% for the children during their school time. Vitamins and minerals will come from a range of fruits and vegetables along within these three major food groups, including 3 serving of vegetable and 2 serving of fruits.

Simultaneously physical activity pattern was analyzed based on data from 24 hour physical activities by children. There were 17 listed physical activities and games questions to assess their frequency of activity on a day.

Under aim 1, investigators were designed a "Healthy Tiffin Box" intervention for children. We were provided a specially designed Tiffin box that will contain five different compartments of various sizes for stuffing with five different food types in order to ensure healthy balanced diet. It was recommended to parents to provide food from all food groups and make a 'Healthy Tiffin Box' with an amount adjusted to the recommended size of the designated compartment. We were suggested a seasonally available and culturally appropriate list of healthy foods and recipes for children. The use of 'Healthy Tiffin Box' was demonstrated to parents, children and school authority by study staff and the benefit of the box will be explained to understand the importance of healthy eating and physical activity practice from their early life.

To achieve specific aim 2, a healthy Tiffin box (intervention material) and healthy eating and active living intervention guideline (intervention module) were developed to deliver healthy lifestyle message encouraging healthy dietary habit and physical activity pattern in order to control childhood overweight and obesity. The guideline was consisted of detail description of healthy dietary behaviour and appropriate physical activity within school environments. There were some pictorial messages and food items in the guideline for clear understanding. We were delivered messages through one hour interactive group session consisting of child and parents pair based on guideline.

Investigators were provided specially designated healthy tiffin box to encourage children healthy eating habit started from their school time. In this feasibility study, children were selected for tiffin box intervention based on their higher BMI and based on consent from their parents. For children aged 11-12 years old, we were collected their assent beside their parent's consent. The tiffin box was designated based on available design of box with addition compartment from the local market. In order to building a healthy tiffin box, we were designed additional four compartments with appropriate portion size for whole grain, snakes, fruits and vegetable. For assessing feasibility of implementing "Healthy Tiffin Box" intervention we were adopted three steps.

* Step 1: Demonstration sessions on healthy Tiffin box and guidelines for children and parents
* Step 2: Implementation of intervention and follow-up
* Step 3: Assessment of intervention among children

Step 1: Investigators were demonstrate to parents and children how they will use healthy Tiffin box for school meal and how healthy eating guideline will guide them to prefer healthy foods with appropriate portion size for their children through group session. We were suggested the parents a list of healthy food items for each compartment of the Tiffin box. Selected parents and children were rigorously trained on healthy eating and active living guideline. We were conducted session with child and mother in pair and give an overview on the following topics related to energy intake and expenditure 1) a decrease in the consumption of unhealthy diets 2) Culturally and seasonally available healthy foods for children 3) proper method of providing food for school 4) increasing the ratio of healthy to unhealthy snacks importance of physical activity during childhood 5) Type of indoor and outdoor activities for children 6) a reduction in screen-based activities.

The training was included interactive lecture on the above topics within children's appropriate time (during Tiffin period or after school time) and demonstration on the proper use of healthy Tiffin box. We were involved children and parents prioritizing few photographs of available healthy and unhealthy foods as first activity; the second activity was involved sorting few existing photographs of active and sedentary, indoor and outdoor activities, and discussion around a photograph of an overweight adolescent boy and girl playing basketball was third activity. Photographs were collected from existing sources through relevant website to understand and encourage discussion amongst children that previously have been shown to be an effective method (Curtin, 2001). We were performed an hour session among school teachers for their understanding about the programme and guideline. As teachers are responsible for children's school hour's activities, they were also be included in the training session.

Step 2: This step was included implementation of intervention and follow-up. We were set goals during the training session on Tiffin box and guideline with the parents and children's. We were asked the parents to provide locally available healthy foods and tasty recopies for their children from all food groups that they have learnt from their session. Parents were also being asked to monitor active physical game during their leisure time. For activities during school, teachers were being requested to reinforce their pupils for physical activity. Selected participants were followed up each weekly by a staff in order to ensure compliance to intervention by providing recommended healthy foods and ensure activities to keep energy balance. Throughout the programme the children and parents were encouraged to find acceptable activity and dietary replacements from available list to ensure healthy energy balance. Teachers were asked to follow children's daily eating patterns as well as physical activity. Our study staffs were followed up each participant weekly up to 4 weeks after the training session and document findings through a check-list.

Step 3: Investigators were assess the feasibility of the intervention among children at the schools. Parents of the students were asked about the intervention to assess compliance. We were developed an assessment tool based on guideline in order to understand problem parents faced while implementing the intervention. This assessment tool (check-list) was used to understand the feasibility of intervention which was consist of prescribed information on diet and physical activity that have been given during training session. The assessments of feasibility of intervention among child and parents pair were conducted in school.

In order to achieve specific aim 3, Investigators were adopted qualitative approach to assess the feasibility of proposed Healthy Tiffin Box intervention for children with higher than a normal BMI for promoting healthy eating and active living in school setting.

Focus group discussion of parents Focus group discussion of children and parents were used to assess the likelihood and acceptance of the proposed future healthy eating and active living intervention as well as their opportunity and barrier to implement such intervention in school setting.

All activities were designed to allow spontaneous discussion amongst the children; the one research officer was act as a facilitator. During focus group discussion, one research officer was responsible for keeping a written record that was include notation of children's responses, relevant quotes, and facilitator observations. An observer was also be present while discussion to observe whether the discussion is continuing according to discussion guideline.

Key Informant interviews (KII) of teachers and policy makers:

Investigators were perform key informant interviews to collect information from a wide range of experts-including teacher and policy makers, involve with schools, planner of schools and parents/guardian- who have detailed knowledge about opportunity of school facilities and experiencing barriers for school health programs. Through these interviews, with their particular knowledge and understanding, Investigators would be able to evaluate insight on nature of the problem and take recommendations for solutions.

ELIGIBILITY:
Inclusion Criteria:

* 2 English medium school and 2 Bengali medium school
* Schools situated at Dhaka North City Corporation.
* Participants both male and female.
* Must be student of grade 3 to grade 9.
* Who will agree to give consent.
* Who have higher than normal BMI, overweight and obese.

Exclusion Criteria:

* Who have normal BMI.
* Who will not agree to give consent.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 831 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Retention rate | 6 months
  No of participant attend in the implementation program on healthy eating and active living and use healthy tiffin box
  * Proportion of children measured for weight
  * Proportion of children measured for height
  * Proportion of children selected for intervention
  * Proportion of children participated in the intervention session
  * No of targeted parents trained on guideline in each session
  * Proportion of planned HEAL intervention session that were delivered

SECONDARY OUTCOMES:
2. Number of participant adhere with healthy eating and active living and use healthy tiffin box intervention | 6 months
  No of children adhere with intervention will be assessed by follow up Check-list
Participants' barrier and facilitators for practicing the implemented intervention program | 6 months
  assessed by qualitative guideline thorough Focus Group Discussion and In depth interview

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Pervin, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No